CLINICAL TRIAL: NCT04525495
Title: Pharmacokinetic and Pharmacodynamic Study of Sildenafil in Neonates and Preterm Infants
Brief Title: Dopamine in Neonate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPMSNUH
Record Dates: First submitted 2020-07-26; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-07

CONDITIONS: Neonates and Preterm Infants
MeSH Terms: interventions — Dopamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dopamine treatment (Experimental)
  Interventions: Drug: Dopamine

INTERVENTIONS:
Drug: Dopamine — Dopamine treatment

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and pharmacodynamics of dopamine which is used as treatment of hypotension in neonate and preterm infant.

ELIGIBILITY:
Inclusion Criteria:

* Admitted at NICU in Seoul National University Hospital, Seoul Asan Hospital or Severance Hospital
* Infants who were diagnosed with hypotension

Exclusion Criteria:

* Congenital heart disease
* Chromosomal anomaly
* Treated with ECMO or CRRT
* Arrhythmia
* Hypovolemic state

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Steady state concentration of dopamine (Css) at 2mcg/kg/min | After continuous infusion for more than 30 minutes at 2mcg/kg/min
  dopamine drug level in blood
Steady state concentration of dopamine (Css) at 5mcg/kg/min | After continuous infusion for more than 30 minutes at 5mcg/kg/min
  dopamine drug level in blood
Steady state concentration of dopamine (Css) at 10mcg/kg/min | After continuous infusion for more than 30 minutes at 10mcg/kg/min
  dopamine drug level in blood
Steady state concentration of dopamine (Css) at 15mcg/kg/min | After continuous infusion for more than 30 minutes at 15mcg/kg/min
  dopamine drug level in blood
Steady state concentration of dopamine (Css) at 20mcg/kg/min | After continuous infusion for more than 30 minutes at 20mcg/kg/min
  dopamine drug level in blood

SECONDARY OUTCOMES:
Blood pressure in mmHg at 2mcg/kg/min | After continuous infusion for more than 30 minutes at 2mcg/kg/min
  Systolic, diastolic and mean blood pressure in mmHg
Blood pressure in mmHg at 5mcg/kg/min | After continuous infusion for more than 30 minutes at 5mcg/kg/min
  Systolic, diastolic and mean blood pressure in mmHg
Blood pressure in mmHg at 10mcg/kg/min | After continuous infusion for more than 30 minutes at 10mcg/kg/min
  Systolic, diastolic and mean blood pressure in mmHg
Blood pressure in mmHg at 10mcg/kg/min | After continuous infusion for more than 30 minutes at 20mcg/kg/min
  Systolic, diastolic and mean blood pressure in mmHg
Heart rate | After continuous infusion for more than 30 minutes at 2mcg/kg/min
Heart rate | After continuous infusion for more than 30 minutes at 5mcg/kg/min
Heart rate | After continuous infusion for more than 30 minutes at 10mcg/kg/min
Heart rate | After continuous infusion for more than 30 minutes at 15mcg/kg/min
Heart rate | After continuous infusion for more than 30 minutes at 20mcg/kg/min
Ejection fraction from Echocardiography | After continuous infusion for more than 30 minutes at 2mcg/kg/min
Ejection fraction from Echocardiography | After continuous infusion for more than 30 minutes at 5mcg/kg/min
Ejection fraction from Echocardiography | After continuous infusion for more than 30 minutes at 10mcg/kg/min
Ejection fraction from Echocardiography | After continuous infusion for more than 30 minutes at 15mcg/kg/min
Ejection fraction from Echocardiography | After continuous infusion for more than 30 minutes at 20mcg/kg/min
Fractional shortening from Echocardiography | After continuous infusion for more than 30 minutes at 2mcg/kg/min
Fractional shortening from Echocardiography | After continuous infusion for more than 30 minutes at 5mcg/kg/min
Fractional shortening from Echocardiography | After continuous infusion for more than 30 minutes at 10mcg/kg/min
Fractional shortening from Echocardiography | After continuous infusion for more than 30 minutes at 15mcg/kg/min
Fractional shortening from Echocardiography | After continuous infusion for more than 30 minutes at 20mcg/kg/min
Tei index from Echocardiography | After continuous infusion for more than 30 minutes at 2mcg/kg/min
  (Mitral valve closure to opening time(ms)-LV ejection time(ms))/LV ejection time(ms)
Tei index from Echocardiography | After continuous infusion for more than 30 minutes at 5mcg/kg/min
  (Mitral valve closure to opening time(ms)-LV ejection time(ms))/LV ejection time(ms)
Tei index from Echocardiography | After continuous infusion for more than 30 minutes at 10mcg/kg/min
  (Mitral valve closure to opening time(ms)-LV ejection time(ms))/LV ejection time(ms)
Tei index from Echocardiography | After continuous infusion for more than 30 minutes at 15mcg/kg/min
  (Mitral valve closure to opening time(ms)-LV ejection time(ms))/LV ejection time(ms)
Tei index from Echocardiography | After continuous infusion for more than 30 minutes at 20mcg/kg/min
  (Mitral valve closure to opening time(ms)-LV ejection time(ms))/LV ejection time(ms)
VTI (velocity time integral) from Echocardiography | After continuous infusion for more than 30 minutes at 2mcg/kg/min
  the area within the spectral curve and indicates how far blood travels during the flow period
VTI (velocity time integral) from Echocardiography | After continuous infusion for more than 30 minutes at 5mcg/kg/min
  the area within the spectral curve and indicates how far blood travels during the flow period
VTI (velocity time integral) from Echocardiography | After continuous infusion for more than 30 minutes at 10mcg/kg/min
  the area within the spectral curve and indicates how far blood travels during the flow period
VTI (velocity time integral) from Echocardiography | After continuous infusion for more than 30 minutes at 15mcg/kg/min
  the area within the spectral curve and indicates how far blood travels during the flow period
VTI (velocity time integral) from Echocardiography | After continuous infusion for more than 30 minutes at 20mcg/kg/min
  the area within the spectral curve and indicates how far blood travels during the flow period

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea